CLINICAL TRIAL: NCT01432106
Title: A Randomized, Double Blind, Active Comparator, Parallel-group Study to Determine Whether the Combination of Valsartan and Aliskiren Provides Cardioprotection in African American Patients With Hypertension and Elements of the Metabolic Syndrome
Brief Title: The Study of Novel Dual Renin Angiotensin Aldosterone System (RAAS) Blockade; Valsartan/Aliskiren in African American Patients With Hypertension and the Metabolic Syndrome
Acronym: SAAVE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Novartis terminated all projects involving aliskiren. Findings of the DMC overseeing the ALTITUDE clinical trial found a higher incidence of adverse events.
Sponsor: University of Michigan (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Kenneth A. Jamerson, Professor of Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPP100AUS20T
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2013-11-18 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension; Metabolic Syndrome
Keywords: Hypertension; Metabolic Syndrome; African American
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — Valsartan; aliskiren; Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aliskiren/Valsartan (Valturna) (Active Comparator): Valturna contains two prescription medicines in one tablet that work together to lower blood pressure. It contains aliskerin (Tekturna), a direct rennin inhibitor (DRI), and valsartan (Diovan), an angiotensin II receptor blocker (ARB). Aliskerin reduces the effect of rennin, and the harmful process that narrows blood vessels. It also helps blood vessels relax and widen so blood pressure is lower. Valsartan can help lower blood pressure by blocking a potent chemical, angiotensin II, which leads to blood vessel constriction and narrowing.
  Interventions: Drug: Aliskerin/Valsartan and Rampiril
- Ramipril (Active Comparator): Ramipril (Altace) is an angiotensin-converting enzyme inhibitor (ACEI). It is a chemical compound that helps create a protein named angiotensin II. Angiotensin II can raise blood pressure by causing your blood vessels to narrow. Altace helps lower blood pressure by decreasing the amount of ACE the body makes. Ramipril has been proven by the investigators to stabilize decline in kidney function in African American patients with evidence of damage.
  Interventions: Drug: Aliskerin/Valsartan and Rampiril

INTERVENTIONS:
Drug: Aliskerin/Valsartan and Rampiril — Patients will start on low dose Ramipril 10 mg or Valturna 150/160 at visit 2, and up-titrate to target dose of Ramipril 20 mg or Valturna 300/320 at visit 3. At visit 5, the addition of Hydrochlorothiazide (HCTZ) or amlodipine will be allowed to achieve the SBP target of < 140 mmHg. High dose will then be maintained throughout the remainder of the study. In case of symptoms of low blood pressures, the study medication may be decreased to the low dose.
  (However, all non-study medication will be manipulated, initially.)
  Other Names: Tekturna (Aliskerin); Diovan (Valsartan); Valturna (Aliskerin/Valsartan; Altace (Ramipril)

SUMMARY:
Study purpose: African Americans with hypertension and markers of metabolic syndrome (small elevations in blood glucose, triglycerides and or weight) are at a high risk of cardiovascular (heart and blood vessel) problems. There is a circulating factor called angiotensin II that increases risk and may be more important in African Americans who have up to 20 times greater risk of losing kidney function and requiring dialysis. Research Investigators, including those at the University of Michigan, found one drug (Ramipril) that blocks angiotensin II effects significantly and improves kidney function in African Americans.

The purpose of The SAAVE Study is to determine whether the combination of two new blockers (Valsartan and Aliskiren) of angiotensin II, are better able to lower blood pressure, also improve some of the risk factors for cardiovascular problems and provide greater protection to the heart and kidneys.

DETAILED DESCRIPTION:
The specific hypothesis of this proposal is that the combination of Valsartan/Aliskiren will provide incremental reduction in blood pressure when compared to traditional blockade of Renin Angiotensin Aldosterone System (RAAS) with ramipril. As an exploratory analysis, we propose that the blood pressure effect will be associated with suppressing plasma aldosterone levels, preserving the availability of nitric oxide, and preventing the development of insulin resistance. Other variables of interest include changes from baseline in adiponectin, Procollagen 1 and 3, osteopontin, cystatin C, and serum K+. In a nested cohort we will determine the impact of novel dual RAAS blockade on left ventricular remodeling.

Should our hypotheses be proven correct and novel dual RAAS blockade is more effective than ramipril in reducing blood pressure, plasma aldosterone, preserving the availability of nitric oxide, as reflected by an increase in asymmetric dimethly arginine (ADMA) levels, and improves cardiovascular remodeling, this would have important implications for the long term prevention of target organ damage and cardiovascular events in this high risk ethnic group.

ELIGIBILITY:
Inclusion Criteria:

1. African American men or women 18 - 80 years of age.
2. Appropriate therapy for high blood pressure consisting of no more than 2 antihypertensives.
3. Patients with at least one marker of Metabolic Syndrome as evidenced by:

   * HDL cholesterol < 35mg/dl (men); < 45 mg/dl (women)
   * Triglycerides > 200mg/dl
   * Fasting Glucose >100mg/dl
   * Waist Circumference: Men >40 inches (102cm); Women > 35 (88cm)
4. Recent copy of EKG.
5. Women able to become pregnant must use reliable contraception (e.g. hormonal contraception and double-barrier methods) throughout this study and for one week after the end of this study. Post-menopausal or surgically sterile women.

Exclusion Criteria:

1. Uncontrolled hypertension.
2. Organ transplant.
3. Hypersensitivity to any study medications
4. Systolic pressure 170 or higher or Diastolic pressure 110 or higher.
5. Cardiovascular events within last 6 months Stroke, Heart Attack, Stent, or Hospitalization for severe Heart Failure.
6. Serum potassium greater than 5.0
7. Heart block without a pacemaker, continuing arrhythmia or valvular heart disease.
8. Blocked renal artery.
9. Patients with severe renal impairment (creatinine 1.7 mg/dl for women and 2.0 mg/dl for men and or estimated GFR <30 mL/min) a history of dialysis, nephritic syndrome, or reno-vascular hypertension.
10. Any condition that may alter medication absorption.
11. Any condition that may place patient at higher risk from participating in study or will jeopardize the evaluation of efficacy or safety.
12. Use of any investigational study medications within 30 days of enrollment
13. Persons unwilling or unable to take regular medications or comply with study protocol.
14. Pregnant or nursing (lactating) women, or women of childbearing potential (defined as all women physiologically capable of becoming pregnant) who do not use reliable methods of contraception: surgical sterilization, bilateral tubal ligation, hormonal contraception, implantable and oral) and double barrier methods if accepted by local regulatory authority and ethics committee. Reliable contraception should be maintained throughout the study and for 7 days after study drug discontinuation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Mean Change in SBP from baseline to 10 weeks (2 weeks on initial dose & 6 weeks on higher dose) | 2 weeks on initial dose & 6 weeks on higher dose

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Jamerson, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States